CLINICAL TRIAL: NCT06920680
Title: ColoReg: A Register for Gastrointestinal Endoscopy Reports and Examination Videos
Status: Recruiting | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Robert Bosch Medical Center (Other); Krankenhaus Barmherzige Brüder, Regensburg (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Klinikum Ludwigsburg (Other)
Responsible Party: Sponsor
Other Study IDs: 151/23-sc
Record Dates: First submitted 2024-09-08; First posted 2025-04-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer; Colonoscopy; Polypectomy
Keywords: colorectal cancer; colonoscopy; standardized documentation; interventional endoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colonoscopy: All patients recruited in a study center are included.

SUMMARY:
With the participants help, the investigators aim to track treatment methods, treatment outcomes, and adverse events, as well as document the treatment strategies used during endoscopic colorectal cancer prevention and treatment. This will allow us to verify if the results from targeted clinical studies and current scientific knowledge are also reflected in the real world. Additionally, the investigators want to use the collected videos and findings to support the training of doctors. During each examination, doctors must be able to accurately assess the inside of the body. Teaching materials for this purpose are scarcely available, often outdated (especially images), and usually show obvious cases. The investigators aim to provide doctors with the opportunity to learn outside of real patient examinations and benefit from the experiences of others.

Furthermore, the investigators want to make the findings and video data accessible to the scientific community. Since scientific studies rarely publish raw data for this purpose, there is currently no large and constantly updated database of findings, images, and videos. If a study requires such data, new data must be collected with great organizational and financial effort. As a result, different studies are only partially comparable, and their significance is reduced.

By publishing the data, a valuable information source for medical professionals in training, continuing education, and advanced training is created. Researchers also benefit from this data: New technologies, such as image analysis software, can be tested and compared on a consistent basis. Therefore, participation in this study makes a valuable contribution to the foundation of good medical care: education, research, and quality assurance.

Primary Study Goal:

The study aims to evaluate the effectiveness and safety of different endoscopic resection techniques. Effectiveness is defined as achieving a complete removal of the lesion (R0 resection) or having a clear follow-up in more than 90% of cases. Safety is defined as having less than 3% of cases result in complications like perforation, uncontrollable bleeding, or the need for unplanned follow-up due to issues like interval bleeding or perforation. The target diagnostic accuracy is 95%.

Secondary Study Goals:

1. Ensure that in 90% of cases, the recommended follow-up interval aligns with current national guidelines based on the number, size, and histopathology of polyps.
2. Achieve successful retrieval of polyps in more than 95% of cases.
3. Document minor bleedings, defined as continuous bleeding for over 30 seconds that requires clipping.

Tertiary Study Goal:

Develop software that can identify and mask sensitive information (such as names, birth dates, examination dates, and video sections outside the human body) in videos from 1,000 examinations, or flag them for manual review. Similarly, the software should identify and remove sensitive text information in the reports, such as names, birth dates, case numbers, examiners, and phone numbers, or mark the text for manual review.

ELIGIBILITY:
Inclusion Criteria:

* Indication for diagnostic or therapeutic colonoscopy

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with planned diagnostic or therapeutic colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 1834 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
R0 Resection Rate by Removal Method (lesion size >= 20 mm) | through study completion, an average of 1 year
  Rate of histologically complete resection for removed pre-cancerous and cancerous lesions >= 20 mm.
Inconspicious follow-up by method of Removal (lesion >= 20 mm) | through study completion, an average of 1 year
  Rate of macroscopically endoscopic follow-up examinations within 1 year if performed
Major Complication Rate (lesion size >= 20 mm) | through study completion, an average of 1 year
  Rate of examination related major complications defined as endoscopically uncontrollable bleedings or perforations.

SECONDARY OUTCOMES:
Intervention time by method of removal (>= 20 mm) | through study completion, an average of 1 year
  Time required from discovery of a polyp to completed treatment including handling of immediate complications.
Rate of unforeseen re-examination within 3 months after polypectomie (lesions >= 20 mm) | through study completion, an average of 1 year
  Rate of unforeseen re-examination within 3 months after polypectomie (lesions >= 20 mm)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Meining, Prof., Study Chair — University Hospital Wuerzburg
Locations (2):
- Germany (2):
  - Robert Bosch Krankenhaus, Stuttgart, Baden-Wurttemberg
  - University Hospital Würzburg, Würzburg, Bavaria

IPD SHARING:
Plan to Share IPD: Yes
Anonymized images from endoscopy examination videos may be published on an research / educational platform.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Study Protocol and ICF will be available at study start. Analytic code will be published after completion of analyses. Individually selected images or video sequences may be anonymously used on a online platform. Due to the experimental nature of this plan no specific time frame is available yet.
Access Criteria: Due to the experimental nature of this plan no specific access criteria are available yet.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT06920680/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT06920680/ICF_001.pdf